CLINICAL TRIAL: NCT03893279
Title: Perception of Smell and Taste During Antibiotic Treatment
Acronym: OGUSTA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0117
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Infectious Disease
MeSH Terms: conditions — Communicable Diseases | interventions — Smell; Taste; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Smell and Taste and questionnaire — The questionnaire must be completed before the antibiotic is taken, if a change of antibiotic is planned (stop of a treatment or addition of another treatment) and at the end of the antibiotic treatment.

SUMMARY:
Antibiotic use may be associated with effects on the perception of smell and taste. These effects are poorly known. The mechanisms can be very diverse, and the effect can be very variable depending on the type of antibiotic used, the dose, and the duration.

The aim of this study is to analyze the perception of the taste and olfactory capacities of patients, during an antibiotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient with bacterial infectious disease requiring antibiotic treatment.
* Having been informed about the study and not having opposed to participate

Exclusion Criteria:

* Patient under legal protection
* Patient refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient meeting the eligibility criteria followed in the department of Infectious and Tropical Diseases of the Croix Rousse Hospital of the Civil Hospitals of Lyon
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Questionnaire on Perception of taste | Time of antibiotic treatment (maximum 6 months)
  Collection of scores on perception of taste, during questionnaires to be completed before, during, and after taking antibiotics.
  Qualitative analysis.
Questionnaire on Perception of smell | Time of antibiotic treatment (maximum 6 months)
  Collection of scores on perception of smell, during questionnaires to be completed before, during, and after taking antibiotics.
  Qualitative analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious and Tropical Diseases of the Croix Rousse Hospital of the Civil Hospitals of Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No